CLINICAL TRIAL: NCT05176899
Title: Real-World Evaluation of Eko Murmur Analysis Software in a Point of Care Setting
Status: Terminated | Type: Observational
Why Stopped: Data collection complete
Sponsor: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021.12
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Murmur, Heart; Innocent Murmurs; Heart Murmurs; Pathologic Murmur
Keywords: artificial intelligence; machine learning
MeSH Terms: conditions — Heart Murmurs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective cohort: Patients who are at least 50 years of age during their primary care exam will undergo SENSORA™ screening if they provide consent.
  Interventions: Device: Use of Eko CORE electronic stethoscope
- Retrospective cohort: Patients who saw participating providers in the 6 months prior to study start date, and who were referred to echocardiogram and/or cardiology, will be included as provider self-control for patient outcomes and referral rates.

INTERVENTIONS:
Device: Use of Eko CORE electronic stethoscope — Recording of heart sounds using electronic stethoscope
  Groups: Prospective cohort

SUMMARY:
The purpose of this research is to evaluate the impact of Eko AI plus EMAS (Eko Murmur Analysis Software) on a clinician's referral decision in a real-world primary care setting. There is an additional objective of understanding patient outcomes when patients are referred for cardiology follow-up and/or echocardiogram.

DETAILED DESCRIPTION:
Eko has developed a platform to aid in screening for cardiac conditions using a digital stethoscope and machine-learning algorithms to detect the presence or absence of heart conditions such as heart murmurs and atrial fibrillation. In June 2022, the US Food and Drug Administration (FDA) granted Eko a 510(k) clearance for the marketing of "Eko Murmur Analysis Software" (EMAS), a set of machine learning algorithms that are able to screen signal quality and identify fundamental heart sounds, distinguish structural murmurs from absent or innocent murmurs, and provide a structural murmur's timing in the cardiac cycle.

This study sets out to evaluate the impact of EMAS on a clinician's referral decision in a real-world primary care setting, with the additional objective of understanding patient outcomes when patients are referred for cardiology follow-up and/or echocardiogram. Providers will receive access to the EMAS screening tool, called the SENSORA™ Disease Detection Platform, which features the FDA cleared 3M™ Littmann® CORE stethoscope paired with the FDA cleared SENSORA™ enterprise application and EMAS AI running on an iPad, which is mounted on a Tryten stand. SENSORA™ will be used by medical assistants or equivalent as part of the initial patient intake process (e.g., during vitals acquisition).

EMAS influence on individual providers will be assessed by reviewing each provider's number of referrals to cardiology and number of echocardiogram orders for the 6 months preceding study start. These values will be compared to cardiac referral and order rates at the end of the study. Patient outcomes data (e.g., cardiology appointment notes, echocardiogram findings, follow up visits scheduled) will be pulled 6 months after the patient is seen by their primary care provider. Secondary objectives include the continued assessment of algorithm performance on a point-of-care population.

ELIGIBILITY:
Inclusion Criteria:

* Patient verbally consents to participation
* Patient is willing to have heart sounds recorded with an electronic stethoscope
* Patient is age 50 years or older

Exclusion Criteria:

* Patient is unwilling or unable to give verbal informed consent
* Patients experiencing a known or suspected acute cardiac event
* Patient is under the age of 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be screened by MedStar study personnel for eligibility from the onsite primary, internal medicine, and geriatric clinics at MedStar. If a patient meets all of the inclusion criteria, and none of the exclusion criteria, they will be approached for participation.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Impact of EMAS on echocardiogram order rates | 01/17/2022 - 11/30/2023
  Echocardiogram order rates before and after SENSORA implementation, for individual providers and aggregated for the site as a whole
Impact of EMAS on cardiologist consult order rates | 01/17/2022 - 11/30/2023
  Cardiology consultation referral rates before and after SENSORA implementation, for individual providers and aggregated for the site as a whole
Impact of EMAS on provider decision-making | 01/17/2022 - 11/30/2023
  Impact of EMAS on provider decision to refer to echocardiogram, cardiologist, or other workup related to cardiac murmur. Measured via a survey administered to each provider after each patient is screened, which asks if SENSORA AI influenced their decision to refer or not to refer. Measured for individual providers and aggregated for the site as a whole.

SECONDARY OUTCOMES:
Impact of EMAS on patient outcomes | 01/17/2022 - 11/30/2023
  VHD discovery rates before and after SENSORA platform implementation, for individual providers and aggregated for the site as a whole
Sensitivity and specificity | 01/17/2022 - 11/30/2023
  EMAS' accuracy (sensitivity and specificity) in detecting structural murmur, compared to an annotator panel

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be de-identified. Data will only be shared with Eko Devices, and not shared with any other researchers.